CLINICAL TRIAL: NCT03200964
Title: Retrospective Analysis of Anesthesia Delivering for Bariatric Surgery
Brief Title: OS Anesthesia Followup of All Bariatric Procedures at One Hospital
Status: Recruiting | Type: Observational
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Jan Mulier, chairman dep anesthesiology, AZ Sint-Jan AV
Other Study IDs: OS bariatric database
Record Dates: First submitted 2017-06-26; First posted 2017-06-27 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Anesthesia Recovery
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: anesthesia given as required for surgical procedure

SUMMARY:
Database registering demographic patient data, anesthesia and surgery information, post operative recovery and complications if any.

DETAILED DESCRIPTION:
Every patient undergoing a bariatric procedure is entered in the data base after the procedure is finished, based on the information available in the medical records.

the study has no end point and keeps collecting data as long as procedures are performed.

The data is analyzed intermittent when medical questions arise on quality and outcome changes due to changes in clinical treatment taken in order to improve individual patient care.

ELIGIBILITY:
Inclusion Criteria:

* all bariatric procedures

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2004-01 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications first month after surgery. | one month followup
  Clavien-Dindoo classification class 2 to 5 used to describe complications

CONTACTS AND LOCATIONS:
Overall Officials: Marco lanckneus, MD, Study Chair — AZ Sint-Jan AV
Locations (1):
- Azsintjan, Bruges, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: publication using data from ongoing registration — https://www.researchgate.net/publication/331811783_Anaesthetic_Factors_Affecting_Outcome_After_Bariatric_Surgery_a_Retrospective_Levelled_Regression_Analysis